CLINICAL TRIAL: NCT04432675
Title: Comparison of the Effects of Crystal Solution (Lactic Acid Ringer's Solution) and Colloid Solution (Hydroxyethyl Starch) on Mother and Fetus After Cesarean Section
Brief Title: Effects of Crystal Solution and Colloid Solution on Mother and Fetus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CINI-AD-20205-13
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2020-06

CONDITIONS: Cesarean Section; Spinal Anesthesia; Parturition
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxyethl starch group (Experimental): 10 ml/kg hydroxyethl starch as well as goal-directed fluid therapy with 3ml/kg hydroxyethl starch
  Interventions: Drug: hydroxyethl starch
- The control group (Active Comparator): 10 ml/kg Lactated Ringer's solution as well as goal-directed fluid therapy with 3ml/kg Lactated Ringer's solution
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: hydroxyethl starch — 10 ml/kg hydroxyethl starch as well as goal-directed fluid therapy with 3ml/kg hydroxyethl starch
  Other Names: Hydroxyethyl Starch 130/0.4 and Sodium Chloride Injection
  Arms: hydroxyethl starch group
Drug: Lactated Ringer's solution — 10 ml/kg Lactated Ringer's solution as well as goal-directed fluid therapy with 3ml/kg Lactated Ringer's solution
  Arms: The control group

SUMMARY:
Comparison of the effects of crystal solution (lactic acid Ringer's solution) and colloid solution (hydroxyethyl starch) on mother and fetus after cesarean section

DETAILED DESCRIPTION:
The Hydroxyethl group use 10 ml/kg hydroxyethl starch as well as goal-directed fluid therapy with 3ml/kg hydroxyethl starch. The control group 10 ml/kg Lactated Ringer's solution as well as goal-directed fluid therapy with 3ml/kg Lactated Ringer's solution. During the whole operation of elective cesarean section

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton pregnancy scheduled for elective cesarean section under CSEA; American Society of Anesthesiologists (ASA) physical status Ⅰ/Ⅱ; Age ranging from 20 to 40 years old.

Exclusion Criteria:

* History of mental disorder or epilepsy; History of central nervous system (CNS) disease; Preexisting or pregnancy-induced hypertension; History of lumber injury; Severe hypovolemia; Allergy or hypersensitivity to norepinephrine; Body mass index (BMI) above 40 kg/m2; Infection at the puncture site; Tricyclic or imipramine antidepressants.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
hypotension | during operation procedure
  The incidence of maternal hypotension during the operation

SECONDARY OUTCOMES:
umbilical vein blood gases | 24 hours
  umbilical vein blood gases
umbilical artery blood gases | 24 hours
  umbilical artery blood gases
Maternal vein blood gase | 24 hours
  Maternal vein blood gase
The incidences of maternal complications | 24 hours
  The incidences of maternal complications such as hypotension, tachycardia, bandycardia, nausea and vomiting, breath difficulty, and dizzy perioperatively.
Hemodynamic data at time point | 24 hours
  Hemodynamic data at time point

CONTACTS AND LOCATIONS:
Overall Officials: Yanghai Cui, Study Chair — China International Neuroscience Institution
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China